CLINICAL TRIAL: NCT01001507
Title: Cluster Randomized Trial of Integration of Family Planning Services Into HIV Care and Treatment in Suba, Kisumu East, Rongo and Migori Districts of Nyanza Province
Brief Title: Integrating Family Planning Services Into HIV Care and Treatment in Nyanza Province, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ibis Reproductive Health (Other); Kenya Medical Research Institute (Other); Tides (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TFR08-02986
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Unintended Pregnancy; HIV Infections
Keywords: Family planning; HIV; Integrated services; Unintended pregnancy; Kenya
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated HIV/FP services (Experimental): Family planning services are integrated into HIV care and treatment services at this facility.
  Interventions: Procedure: Integrated family planning/HIV care and treatment services
- Standard (non-integrated), referral-based, services (No Intervention): Patients from the HIV care and treatment clinic will be referred for family planning services, and will not receive FP services by the HIV care provider

INTERVENTIONS:
Procedure: Integrated family planning/HIV care and treatment services — Family planning services will be provided during the patient's HIV care visit.
  Arms: Integrated HIV/FP services

SUMMARY:
This is a cluster randomized trial comparing the integration of family planning services into HIV care and treatment programs versus the standard referral for family planning services outside of HIV care and treatment programs within Suba, Kisumu East, Rongo and Migori districts in Nyanza province.

DETAILED DESCRIPTION:
The study will have three parts. During the first part (3 months), baseline data on contraceptive prevalence and unintended pregnancy will be collected at 18 PSCs that are supported by the FACES program in Suba, Kisumu East, Nyatike, Rongo and Migori Districts. Also during this first part, information about knowledge, attitudes and practices related to family planning will be obtained from patients and from clinicians at the sites. During the second part (3 months), an intervention consisting of integrating family planning services will be designed and implemented at twelve of the 18 FACES-supported PSCs. We aim to utilize a 2:1 integration:control model, with delayed integration so as to gradually expand the integration of FP and HIV services throughout the 18 sites, while maintaining the ability to test hypotheses on the effects of integration on health outcomes. After collecting the baseline data, we plan to stratify the clinics into two categories based on the overall patient volume and differences in the structure of family planning provision, i.e., whether or not there is a specific MCH division providing family planning at the site or not. Randomization of sites will then occur among clinics in each of these strata, with a ratio of two intervention sites (integrated model) to one control site (family planning provided in the standard manner at the site). During the third and last part (12 months), data on prevalence more effective contraception and unintended pregnancy will be collected from each of the 18 sites. At the end of part three, information about knowledge, attitudes and practices related to family planning again will be obtained from patients and from clinicians at the sites. In addition, we will administer questionnaires assessing the acceptability of family planning services to patients, and in addition clinic staff will be answer a questionnaire assessing the feasibility of providing integrated family planning services. After 12 months of data collection, the 6 control sites were integrated and data were collected for an additional 11 months from all 18 sites to assess the sustainability of the intervention under the Ministry of Health.

The study population will primarily consist of HIV-positive men and non-pregnant, HIV-positive women of reproductive age who obtain care at the FACES-supported PSCs in Suba, Kisumu East, Rongo and Migori Districts in Nyanza Province, Kenya. In addition, study subjects will also include clinic staff at the FACES centers included in the study.

ELIGIBILITY:
Inclusion Criteria:

For health facilities:

* Each site must be providing HIV care and treatment services

For participants:

* Women aged 18-45, not pregnant, HIV+, receiving HIV care at that health facility
* Men aged 18 and above, HIV+, receiving HIV care at that health facility

Exclusion Criteria:

For health facilities

* If they do not meet the inclusion criteria listed above
* If they are already providing integrated comprehensive HIV care and treatment that includes on-site family planning counseling and provision

For participants:

* Participants are excluded if they do not meet the inclusion criteria listed above.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5040 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Prevalence More Effective Contraception (defined as hormonal methods, intrauterine devices, and permanent methods) | 1 year post integration/site initiation and 2 years post integration/site initiation
Pregnancy rate | 1 year post integration/study initiation and 2 years post integration/site initiation

SECONDARY OUTCOMES:
Knowledge of contraceptive methods among HIV-positive women | baseline (months 1-3); post-intervention (months 9-12)
Knowledge of contraceptive methods among providers | baseline (months 1-3); post-intervention (months 9-12)
Acceptability of family planning services | baseline (months 1-3); post-intervention (months 9-12)
Feasibility of providing family planning services at HIV care and treatment centers | months 9-12
Reproductive intentions of HIV-infected women receiving care and treatment | months 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Craig Cohen, MD, MPH, Principal Investigator — University of California, San Francisco; Daniel Grossman, MD, Principal Investigator — Ibis Reproductive Health; Elizabeth Bukusi, MBChB, PhD, Principal Investigator — Kenya Medical Research Institute; Sara Newmann, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Migori District Hospital, Migori, Kenya

REFERENCES:
- [Derived] Cohen CR, Grossman D, Onono M, Blat C, Newmann SJ, Burger RL, Shade SB, Bett N, Bukusi EA. Integration of family planning services into HIV care clinics: Results one year after a cluster randomized controlled trial in Kenya. PLoS One. 2017 Mar 22;12(3):e0172992. doi: 10.1371/journal.pone.0172992. eCollection 2017. PMID 28328966